CLINICAL TRIAL: NCT04031326
Title: Feasibility and Effectiveness of LENA Home in the Every Child Succeeds Home Visiting Program
Brief Title: Randomized Trial of LENA Home in A Home Visiting Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Every Child Succeeds (Unknown); The Carol Ann and Ralph V. Haile, Jr./U.S. Bank Foundation (Unknown); Bethesda, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-8501
Record Dates: First submitted 2019-02-16; First posted 2019-07-24 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2020-06

CONDITIONS: Parent-Child Relations; Language Development
Keywords: home visiting; LENA; infant language development; parenting

STUDY DESIGN:
Intervention Model Description: This is a single-blind randomized trial with 2 groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LENA Home (Experimental): Home visitors assigned to the intervention group will be trained to use and administer LENA Home in addition to the standard ECS curriculum during designated home visits beginning when the child is between 6- and 9-months old.
  Interventions: Behavioral: LENA Home
- Standard Practice (No Intervention): Home visitors assigned to the control group will administer the standard ECS curriculum only

INTERVENTIONS:
Behavioral: LENA Home — LENA Home is a 13-week curriculum designed to add an early-language focus to existing home visiting or parent education programs for children ages birth to three. It employs LENA wearable audio recorder technology and targeted content to help parents and other caregivers increase interactive talk. There are 13 weekly one-on-one sessions, including modules on parent-child reading and increasing verbal interaction during typical home activities. Sessions include videos, practical techniques, and feedback from LENA recordings via intuitive reports to help parents talk more with their children. LENA Home reports provide data on adult words spoken to the child (AWC) and conversational turns (CTC). LENA Home has been shown to increase interactive talk and child language ability and informs parents how much they are talking with their children in an objective way.
  Arms: LENA Home

SUMMARY:
This study evaluates feasibility and efficacy of adding the LENA Home program to the standard Every Child Succeeds (ECS) home visiting curriculum. Half of the participants will receive the standard ECS curriculum during normally scheduled home visits, while the other half will receive this plus LENA Home.

DETAILED DESCRIPTION:
Every Child Succeeds is a program that uses home visiting as a preventive strategy to support low income families in providing stimulating, safe, and nurturing environments for their young children. Most families in home visiting have experienced adversity in their lives, and had inadequate parenting role models as they grew up. Home visitors visit families during pregnancy through the child reaching three years of age, providing information, teaching, and resources to help parents provide the best possible start for their children.

LENA Home is a 13-week curriculum designed to add an early-language focus to existing home visiting or parent education programs for children ages birth to three. It employs LENA wearable audio recorder technology and targeted content to help parents and other caregivers increase interactive talk. There are 13 weekly one-on-one sessions, including modules on parent-child reading and increasing verbal interaction during typical home activities. Sessions include videos, practical techniques, and feedback from LENA recordings via intuitive reports to help parents talk more with their children. LENA Home reports provide data on adult words spoken to the child (AWC) and conversational turns (CTC). LENA Home has been shown to increase interactive talk and child language ability and informs parents how much they are talking with their children in an objective way.

Upon completion of the study, we will have more information regarding whether (1) LENA Home can be successfully integrated into existing home visiting programs (feasibility), (2) children exposed to LENA have larger vocabularies than those who do not receive the intervention, (3) mothers using LENA engage in more literacy-promoting behaviors relative to controls, and (4) LENA improves parent-child interactions (utility).

ELIGIBILITY:
Inclusion Criteria:

1. enrollment in the Every Child Succeeds home visiting program,
2. child age between 6- and 9-months old,
3. English-speaking household,
4. child gestation of at least 32 weeks,
5. child has no known neurobehavioral/genetic syndrome or brain injury likely to cause language delay,
6. maternal age at least 15 years old.

Exclusion Criteria:

Not meeting the above criteria.

Ages: 6 Months to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Absolute Word Count | Baseline, Midpoint (6-7 week visit), Endpoint (13 weeks)
  The LENA Home recording device measures Absolute Word Count (AWC) over an approximately 13-hour recording period at each recording. This outcome will involve change in AWC between baseline and a Midpoint assessment (approximately 6-7 weeks) and Endpoint (13-weeks).
Change in Conversational Turns Count | Baseline, Midpoint (6-7 week visit), Endpoint (13 weeks)
  The LENA Home recording device measures Conversational Turns Count (CTC) over an approximately 13-hour recording period at each recording. This outcome will involve change in CTC between baseline and a Midpoint assessment (approximately 6-7 weeks) and Endpoint (13-weeks).
Change in LENA Snapshot Language Assessment Score | Baseline, Midpoint (6-7 week visit), Endpoint (13 weeks)
  The LENA Developmental Snapshot is a questionnaire that provides parents with an

SECONDARY OUTCOMES:
Change in DialogPR-I/T (shared reading quality) Score | Baseline and Endpoint (13 weeks).
  Dialog PR-I/T is a 10-item measure of shared reading quality (interactivity) for infants and toddlers developed by the PI that is derived from the validated DialogPR measure for older children. It involves evidence-based behaviors such as lap sitting, use of child-directed speech, and verbal responsivity. Range is 0-30, higher score suggests more interactive, nurturing reading.
Change in ScreenQ-I/T (screen-based media use) | Difference in score between Baseline and Endpoint (13 weeks)
  ScreenQ-I/T is a 10-item composite measure of screen-based media use in the home referenced to current AAP guidelines for infants and toddlers, developed by the PI that is based on the validated ScreenQ measure for older children. Range is 0-23 points, higher scores suggest greater use contrary to AAP guidelines and greater developmental/health risk.
Change in StimQ-I (home cognitive environment) | Baseline and Endpoint (13 weeks)
  The StimQ-I is a validated assessment of parent report measure of cognitive stimulation in the home for children up to 18-months old involving 4 subscales: availability of learning materials, parental involvement in developmental advance, parental verbal responsivity, and reading. Higher scores suggest more stimulating parental behaviors.
Change in SPEAK (parenting mindset) score | Baseline and Endpoint (13 weeks)
  The SPEAK assessment is an assessment of parental mindset towards their infant's development. Higher score suggests more empowered parental mindset.

CONTACTS AND LOCATIONS:
Overall Officials: John Hutton, MD MS, Principal Investigator — Assistant Professor
Locations (1):
- Cincinnati Children's Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Access to data will be restricted to protect the privacy of enrolled subjects. It may be made available in a de-identified fashion in the future.

REFERENCES:
- [Background] Bowers K, Folger AT, Zhang N, Sa T, Ehrhardt J, Meinzen-Derr J, Goyal NK, Van Ginkel JB, Ammerman RT. Participation in Home Visitation is Associated with Higher Utilization of Early Intervention. Matern Child Health J. 2018 Apr;22(4):494-500. doi: 10.1007/s10995-017-2415-8. PMID 29388114
- [Background] Donovan EF, Ammerman RT, Besl J, Atherton H, Khoury JC, Altaye M, Putnam FW, Van Ginkel JB. Intensive home visiting is associated with decreased risk of infant death. Pediatrics. 2007 Jun;119(6):1145-51. doi: 10.1542/peds.2006-2411. PMID 17545382
- [Background] Gilkerson J, Richards JA, Warren SF, Oller DK, Russo R, Vohr B. Language Experience in the Second Year of Life and Language Outcomes in Late Childhood. Pediatrics. 2018 Oct;142(4):e20174276. doi: 10.1542/peds.2017-4276. Epub 2018 Sep 10. PMID 30201624
- See also: Related Info — https://www.everychildsucceeds.org/
- See also: Related Info — https://www.lena.org/about/